CLINICAL TRIAL: NCT03311906
Title: Clinical and Laboratory Effect of 0.8% Hyaluronic Acid Gel in Conventional Treatment of Moderate to Severe Chronic Periodontitis
Brief Title: Evaluation of the Efficacy of 0.8% Hyaluronic Acid Gel
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Riyadh Colleges of Dentistry and Pharmacy (Other)
Responsible Party: Principal Investigator, Nour Al Shammari, Senior Resident, Riyadh Colleges of Dentistry and Pharmacy
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: FPGRP/43631003/73
Record Dates: First submitted 2017-10-02; First posted 2017-10-17 (Actual); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Hyaluronic Acid; Tooth Exfoliation; Root Planing

STUDY DESIGN:
Intervention Model Description: A split mouth study design is used where all participants receive both interventions
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Test side (Experimental): Scaling and Root Planing 0.8% Hyaluronic acid gel
  Interventions: Drug: 0.8% Hyaluronic Acid; Procedure: Scaling and Root Planing
- Control Side (Active Comparator): Scaling and Root Planing
  Interventions: Procedure: Scaling and Root Planing

INTERVENTIONS:
Drug: 0.8% Hyaluronic Acid — Application of 0.8% hyaluronic acid after scaling and root planing
  Other Names: Gengigel
  Arms: Test side
Procedure: Scaling and Root Planing — Scaling of the teeth using hand and ultrasonic scalers followed by planing of the root with curettes

SUMMARY:
assess the clinical and laboratory effects of the local and sub gingival application of a 0.8% hyaluronic acid gel (GENGIGEL®) as an adjunct to scaling and root planning (SRP) in chronic moderate to severe periodontitis patients as indicated by expression of Human Beta Definsin-2 (HBD2) in gingival crevicular fluid (GCF).

DETAILED DESCRIPTION:
Patients who fulfilled the selection criteria will be included in the study. One quadrant will be treated with HA gel (test) and the other without to serve as control. Clinical examination will be done in a dental chair under standard conditions of light, using mouth mirror and graduated Williams Periodontal Probe.

All patients will receive full mouth scaling and root planing with hand instruments and ultrasonic scalers at baseline. Thereafter, in the test quadrant, 1 ml of 0.8% hyaluronic acid gel will be administered subgingivally in all selected test sites at baseline and 1 week later. The following clinical parameters will be recorded at baseline, after 6 weeks and 12 weeks post treatment. Oral hygiene instructions will be given to all patients. The clinical measurements and treatment will be performed by a single examiner.For every patient and control subject, GCF samples will be collected at baseline, 6 weeks and 12 weeks post treatment. The samples will be pooled from two periodontal sites with clinical attachment level of 3 mm or more (in the two different quadrants). The sampling area will be isolated with cotton rolls and carefully will be cleaned supragingivally with sterile cotton pellets. A sterile absorbent paper point will be inserted into the gingival crevice or pocket until resistance will be felt. The paper point will be held in place for 30 s and then will be transferred to a vial containing 100 μL of distilled water and vigorously will be mixed. The paper points will be removed, and the samples will be centrifuged and will be washed twice with distilled water. The resultant pellets will be resuspended in 0.4 mL of distilled water. The samples will be coded and stored at -70 °C until use for ELISA test for identification of Human beta Defensin-2.

ELIGIBILITY:
Inclusion Criteria:

* Patients should be systemically healthy with moderate to severe chronic periodontitis of more than 4 mm probing depth in at least two sites in different quadrants.
* Patient should exhibit no known allergies
* Participants should have the ability to attend the hospital regular intervals.

Exclusion Criteria:

* pregnancy
* nursing
* hypertension
* patient with chronic diseases such as diabetes mellitus or rheumatoid arthritis. -Participants should not be under antibiotics and\or had receive any periodontal therapy for the last 6 months.
* Participants should not taking drugs that could affect the state of the gingival tissues.
* Participants must not be undergoing orthodontic therapy, caries free
* Participants must not be using any other supplemental plaque control measures like mouthwashes.
* Participants should not have the habit of taking alcohol, smoking or chewing tobacco and do not suffer from any systemic disease.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2017-10-02 (Actual)

PRIMARY OUTCOMES:
Clinical Attachment Level (CAL) change | baseline, six weeks, 12 weeks
  Distance from the cementoenamel junction to the base of gingival sulcus using a UNC15 probe
Probing Depth change | baseline, six weeks, 12 weeks
  It's the distance from the gingival margin to base of the sulcus
Gingival Index change (Loe and Silness, 1963) | baseline, six weeks, 12 weeks
  To assess the gingival condition and record qualitative chances in the gingiva
Plaque index change (Loe and Silness, 1964) | baseline, six weeks, 12 weeks
  To measure the state of oral hygiene
Papillary Bleeding Index change (Muhlemann, 1977) | baseline, six weeks, 12 weeks
  immediate evaluation of the patient's gingival motivation and condition

SECONDARY OUTCOMES:
HBD-2 change | baseline, six weeks, 12 weeks
  By take gingival crevicular fluid sample elisa test

CONTACTS AND LOCATIONS:
Overall Officials: Sanaa M Shafshak, PhD, Study Director — Riyadh Colleges of Dentistry and Pharmacy
Locations (1):
- Riyadh Colleges of Dentistry and Pharmacy, Riyadh, AlRiyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brogden KA. Antimicrobial peptides: pore formers or metabolic inhibitors in bacteria? Nat Rev Microbiol. 2005 Mar;3(3):238-50. doi: 10.1038/nrmicro1098. PMID 15703760
- [Result] Diamond DL, Kimball JR, Krisanaprakornkit S, Ganz T, Dale BA. Detection of beta-defensins secreted by human oral epithelial cells. J Immunol Methods. 2001 Oct 1;256(1-2):65-76. doi: 10.1016/s0022-1759(01)00442-2. PMID 11516756
- [Result] Embery G, Waddington RJ, Hall RC, Last KS. Connective tissue elements as diagnostic aids in periodontology. Periodontol 2000. 2000 Oct;24:193-214. doi: 10.1034/j.1600-0757.2000.2240109.x. No abstract available. PMID 11276867
- [Result] Garcia JR, Jaumann F, Schulz S, Krause A, Rodriguez-Jimenez J, Forssmann U, Adermann K, Kluver E, Vogelmeier C, Becker D, Hedrich R, Forssmann WG, Bals R. Identification of a novel, multifunctional beta-defensin (human beta-defensin 3) with specific antimicrobial activity. Its interaction with plasma membranes of Xenopus oocytes and the induction of macrophage chemoattraction. Cell Tissue Res. 2001 Nov;306(2):257-64. doi: 10.1007/s004410100433. PMID 11702237
- [Result] Gontiya G, Galgali SR. Effect of hyaluronan on periodontitis: A clinical and histological study. J Indian Soc Periodontol. 2012 Apr;16(2):184-92. doi: 10.4103/0972-124X.99260. PMID 23055583
- [Result] Gorr SU. Antimicrobial peptides in periodontal innate defense. Front Oral Biol. 2012;15:84-98. doi: 10.1159/000329673. Epub 2011 Nov 11. PMID 22142958
- [Result] Gorr SU, Abdolhosseini M. Antimicrobial peptides and periodontal disease. J Clin Periodontol. 2011 Mar;38 Suppl 11:126-41. doi: 10.1111/j.1600-051X.2010.01664.x. PMID 21323710
- [Result] Haffajee AD, Socransky SS. Microbial etiological agents of destructive periodontal diseases. Periodontol 2000. 1994 Jun;5:78-111. doi: 10.1111/j.1600-0757.1994.tb00020.x. No abstract available. PMID 9673164
- [Result] Heitz-Mayfield LJ. How effective is surgical therapy compared with nonsurgical debridement? Periodontol 2000. 2005;37:72-87. doi: 10.1111/j.1600-0757.2004.03797.x. No abstract available. PMID 15655026
- [Result] Jentsch H, Pomowski R, Kundt G, Gocke R. Treatment of gingivitis with hyaluronan. J Clin Periodontol. 2003 Feb;30(2):159-64. doi: 10.1034/j.1600-051x.2003.300203.x. PMID 12622859
- [Result] Johannsen A, Tellefsen M, Wikesjo U, Johannsen G. Local delivery of hyaluronan as an adjunct to scaling and root planing in the treatment of chronic periodontitis. J Periodontol. 2009 Sep;80(9):1493-7. doi: 10.1902/jop.2009.090128. PMID 19722800
- [Result] Loe H. The Gingival Index, the Plaque Index and the Retention Index Systems. J Periodontol. 1967 Nov-Dec;38(6):Suppl:610-6. doi: 10.1902/jop.1967.38.6.610. No abstract available. PMID 5237684
- [Result] LOE H, SILNESS J. PERIODONTAL DISEASE IN PREGNANCY. I. PREVALENCE AND SEVERITY. Acta Odontol Scand. 1963 Dec;21:533-51. doi: 10.3109/00016356309011240. No abstract available. PMID 14121956
- [Result] Moseley R, Waddington RJ, Embery G. Hyaluronan and its potential role in periodontal healing. Dent Update. 2002 Apr;29(3):144-8. doi: 10.12968/denu.2002.29.3.144. PMID 11989392
- [Result] Muhlemann HR. Psychological and chemical mediators of gingival health. J Prev Dent. 1977 Jul-Aug;4(4):6-17. No abstract available. PMID 275483
- [Result] Niyonsaba F, Ushio H, Nakano N, Ng W, Sayama K, Hashimoto K, Nagaoka I, Okumura K, Ogawa H. Antimicrobial peptides human beta-defensins stimulate epidermal keratinocyte migration, proliferation and production of proinflammatory cytokines and chemokines. J Invest Dermatol. 2007 Mar;127(3):594-604. doi: 10.1038/sj.jid.5700599. Epub 2006 Oct 19. PMID 17068477
- [Result] Pereira AL, Franco GC, Cortelli SC, Aquino DR, Costa FO, Raslan SA, Cortelli JR. Influence of periodontal status and periodontopathogens on levels of oral human beta-defensin-2 in saliva. J Periodontol. 2013 Oct;84(10):1445-53. doi: 10.1902/jop.2012.120321. Epub 2012 Nov 23. PMID 23173827
- [Result] Pilloni A, Annibali S, Dominici F, Di Paolo C, Papa M, Cassini MA, Polimeni A. Evaluation of the efficacy of an hyaluronic acid-based biogel on periodontal clinical parameters. A randomized-controlled clinical pilot study. Ann Stomatol (Roma). 2011 Mar;2(3-4):3-9. Epub 2012 Jan 27. PMID 22545183
- [Result] Pirnazar P, Wolinsky L, Nachnani S, Haake S, Pilloni A, Bernard GW. Bacteriostatic effects of hyaluronic acid. J Periodontol. 1999 Apr;70(4):370-4. doi: 10.1902/jop.1999.70.4.370. PMID 10328647
- [Result] Polepalle T, Srinivas M, Swamy N, Aluru S, Chakrapani S, Chowdary BA. Local delivery of hyaluronan 0.8% as an adjunct to scaling and root planing in the treatment of chronic periodontitis: A clinical and microbiological study. J Indian Soc Periodontol. 2015 Jan-Feb;19(1):37-42. doi: 10.4103/0972-124X.145807. PMID 25810591
- [Result] Porter EM, Liu L, Oren A, Anton PA, Ganz T. Localization of human intestinal defensin 5 in Paneth cell granules. Infect Immun. 1997 Jun;65(6):2389-95. doi: 10.1128/iai.65.6.2389-2395.1997. PMID 9169779
- [Result] Xu Y, Hofling K, Fimmers R, Frentzen M, Jervoe-Storm PM. Clinical and microbiological effects of topical subgingival application of hyaluronic acid gel adjunctive to scaling and root planing in the treatment of chronic periodontitis. J Periodontol. 2004 Aug;75(8):1114-8. doi: 10.1902/jop.2004.75.8.1114. PMID 15455740